CLINICAL TRIAL: NCT00763425
Title: Prospective Randomized Comparison of Cold Snare Polypectomy and Conventional Polypectomy
Acronym: COLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Showa Inan General Hospital (Other)
Responsible Party: Principal Investigator, Akira Horiuchi, Digestive Disease Center, Showa Inan General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200888
Record Dates: First submitted 2008-09-29; First posted 2008-10-01 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Colorectal Cancer
Keywords: polypectomy; colonic polyp; colorectal polyp; colorectal cancer prevention
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Procedure: cold polypectomy
- 2 (Active Comparator)
  Interventions: Procedure: conventional polypectomy

INTERVENTIONS:
Procedure: cold polypectomy — The removal of small colorectal polyps up to 8 mm is performed using cold snare polypectomy.
  Other Names: cold snare polypectomy
  Arms: 1
Procedure: conventional polypectomy — The removal of small colorectal polyps up to 8 mm is performed using conventional polypectomy.
  Other Names: polypectomy
  Arms: 2

SUMMARY:
The aim of this study is to compare cold snare polypectomy and conventional polypectomy for the removal and retrieval of small colorectal polyps.

Cold snare polypectomy for colorectal polyps up to 8 mm is expected to be more effective than conventional polypectomy.

ELIGIBILITY:
Inclusion criteria:

* Men or women between 20 and 100 years of age

Exclusion Criteria:

* Exclusion criteria include age less than 20 years old
* Pregnant, American Society of Anesthesiologists class III and IV
* Overweight (body weight > 100 kg)
* Allergic to the drugs used or its components (soybeans or eggs)
* Poor bowel preparation or post-colorectal surgery.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-09; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Complete removal rate of colorectal polyps | two weeks after each polypectomy

SECONDARY OUTCOMES:
Complication rate | two weeks after each polypectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Showa Inan General hospital, Komagane, Nagano, Japan